CLINICAL TRIAL: NCT01004120
Title: Double-blind, Placebo Controlled, Randomised, Cross-over Study to Determine the Effect of a Prebiotic Galactooligosaccharide on Microbiota and Metabolic Syndrome Risk Factors in Overweight Adults
Brief Title: Efficacy of a Prebiotic Galactooligosaccharide to Reduce Metabolic Syndrome Risk Factors in Overweight Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clasado (Industry)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: COMSE
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome | interventions — 4'-galactooligosaccharide; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MDn (Placebo Comparator)
  Interventions: Dietary Supplement: Maltodextrin
- B-GOS (Active Comparator)
  Interventions: Dietary Supplement: Bimuno

INTERVENTIONS:
Dietary Supplement: Bimuno — 5.5g daily intake
  Other Names: Galactooligosaccharide
  Arms: B-GOS
Dietary Supplement: Maltodextrin — 5.5g daily intake
  Other Names: Dexrins
  Arms: MDn

SUMMARY:
The traditional risk factors for obesity are inappropriate diet, lack of exercise and genetic factors. However, recent observations have involved gut microbiota profiles as having an additional influence. In this case, there exists the possibility to modulate this through diet. Research has shown that the gut microbiota of both obese humans and mouse models of obesity is altered towards less beneficial one compared to lean counterparts. This raises the possibility of modulating the gut microbiota as a novel strategy in tackling the epidemic of obesity and diabetes sweeping the developed world. In addition, a more direct effect of high-fat induced disruption of the intestinal microbiota has also been seen with a murine model. Elevated circulating levels of lipopolysaccharide (LPS) a major building block and antigen of Gram-negative bacteria, was shown to generate a low grade chronic inflammation, termed metabolic endotoxemia, which then onsets insulin resistance. High-fat diets were shown to disrupt the Gram-negative intestinal populations of these animals, liberating LPS. The effects of prebiotics on the microbiota or metabolic syndrome (combination of disorders that increase the risk of developing cardiovascular disease and diabetes) in overweight adults have not been investigated thus far. The investigators therefore propose to investigate the effect of galactooligosaccharide (GOS) on the faecal microbiota and metabolic syndrome risk factors in overweight adults in a double-blind, randomised, placebo controlled, cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* 18-65y
* BMI >25 kg/m2

Exclusion Criteria:

* Suffered from a myocardial infarction/stroke or cancer in the past 12 months
* Diabetic or suffering from endocrine disorders
* Suffer from renal or bowel disease/gut disorder or have a history of cholestatic jaundice or pancreatitis
* Requirements to take long-term medication for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* History of alcohol or drug abuse
* Planning or on a weight reducing regime
* Taking antioxidant (or phytochemical), probiotic or prebiotics supplements
* Pregnant or lactating women or those planning pregnancy in the next 6 months or of child-bearing age who are not using contraception
* Use of antibiotics within the previous 1 month
* Anemic
* Smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Faecal microbiota changes enumerated by Fluorescent In Situ Hybridisation and qualitatively assessed by Denaturing Gradient Gel Electrophoresis. | 3 months
Lipid profile (total, LDL and HDL cholesterol, triglycerides and non-esterified fatty acids) | 3 months
Inflammatory/thrombotic biomarkers (including C-reactive protein, TNF-a, IL6, IL-8, IL-10, sCD40L, sP-selectin, t-PA) | 3 months

SECONDARY OUTCOMES:
Insulin resistance derived from fasted measures of glucose and insulin ratio | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jelena Vulevic, PhD, Principal Investigator — The University of Reading
Locations (1):
- School of Chemistry, Food Biosciences and Pharmacy, The University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Vulevic J, Juric A, Tzortzis G, Gibson GR. A mixture of trans-galactooligosaccharides reduces markers of metabolic syndrome and modulates the fecal microbiota and immune function of overweight adults. J Nutr. 2013 Mar;143(3):324-31. doi: 10.3945/jn.112.166132. Epub 2013 Jan 9. PMID 23303873